CLINICAL TRIAL: NCT06902337
Title: Gender Differences in Gastric Cancer Care and Its Adherence to Guidelines in Germany: A Observational Retrospective Cohort Study With Administrative Routine and Cancer Registry Data From 2017-2021
Brief Title: Gender Differences in Gastric Cancer Care and Its Adherence to Guidelines in Germany
Acronym: MaGen
Status: Active, not recruiting | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Principal Investigator, Rene Mantke, MD, PhD, Head of Surgery at University Hospital Brandenburg an der Havel, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: MaGen (01VSF24051); 01VSF24051 (Other Grant/Funding Number: Innovation Fund of the Federal Joint Committee, Germany)
Record Dates: First submitted 2025-03-21; First posted 2025-03-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric cancer; Sex differences; Clinicopathological characteristics; Treatment; Mortality; Survival; Treatment guidelines; Administrative routine data; Cancer registry data
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with gastric adenocarcinoma: Gastric carcinoma (ICD-10-GM C16) Patients with gastric carcinoma in the years 2017-2021 in Germany, minimum age 18 years

SUMMARY:
Background: Gastric cancer is the fifth most common cancer globally and the fourth leading cause of cancer-related mortality. While gender differences in gastric cancer care are underexplored in Germany, international studies have revealed disparities in aspects such as histology, co-morbidities, treatment approaches, and survival outcomes. This study aims to explore gender-specific variations in clinical management and their impact on mortality, complications, and survival rates in gastric carcinoma patients in Germany.

Methods: This nationwide, retrospective cohort study will analyze data from the German Diagnosis-Related Group statistic and regional clinical cancer registries from 2017 to 2021. The study will evaluate both datasets separately, providing a comprehensive view of gender differences in gastric cancer care. Primary outcomes include hospital mortality and survival rates, while secondary endpoints include surgical complications, treatment modalities, and postoperative outcomes. The analysis will investigate whether gender influences tumor characteristics, access to treatment, and therapy effectiveness. Statistical methods such as descriptive analysis, regression models, and survival analysis will be applied to identify gender-related variations in diagnosis, treatment, and outcomes.

Discussion: By identifying potential gender disparities in diagnosis, treatment, and outcomes, the findings may inform revisions to clinical guidelines and support the development of more personalized treatment strategies. This study aims to improve the quality of care for gastric cancer patients and promote more individualized, sex-sensitive medical practices.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common cancer globally and the fourth leading cause of cancer-related mortality. While there is a lack of current data on gender differences in gastric cancer care in Germany, several international studies conducted on the basis of clinical cancer registry data have pointed to the relevance of this aspect in recent years. The analyses showed significant differences between women and men in aspects such as histology, co-morbidities, operations and therapies performed, and survival rates.

In Germany in 2017, 15,690 people were diagnosed with gastric cancer, of which 6190 were women (39%) and 9490 men (61%). The age-standardized rate of new cases is 7.8 for women and 14.9 for men. The risk of developing the disease increases with age in both sexes; men develop stomach cancer on average at the age of 71 and women at 76 years of age. There are regional differences between the federal states of Germany in all key figures. For example, in the state of Bavaria in 2019, both sexes have an above-average 5-year survival rate of 46.1% for men and 50.7% for women, while in the state of Brandenburg there is a large difference in this ratio between men (38.5%) and women (46.0%).

With regard to hospital mortality in Germany, an analysis of data from the DRG statistics for the years 2009 -2015 showed that the highest mortality rate of 11.7% was observed in patients undergoing visceral surgery in complex gastric surgery (in comparison, average hospital mortality among patients undergoing visceral surgery: 1.9%).

The aim of the project is to use routine data of the DRG statistic and data from the clinical cancer registries of the federal states to determine whether there are differences between women and men in the clinical care of gastric carcinomas and whether such different care has an impact on the mortality rate, complications and survival time of those affected.

Data from the hospital statistics (DRG statistics) and data from the clinical cancer registries are used as the data basis for the above-mentioned research questions and evaluated separately from each other.

In a first step, it will be investigated whether and to what extent women and men already differ in tumor characteristics (diagnosis, localization, histology, UICC stage, etc.) and in possible co-morbidities and co-variates such as age.

In a second step, the therapy (surgical procedures, oncological therapies) is analyzed under the focus variable gender. The aim here is to analyze whether women and men receive the same therapies if, for example, the tumor characteristics have the same tumor characteristics, or whether there are differences in both access and type of therapies.

In a third step, both the influence of the tumor characteristics and the therapies used on the outcome of the therapies will be investigated under gender-specific aspects. These include, for example, complications after surgery, side effects of oncological therapies, length of hospital stay, hospital mortality or long-term survival. It is of particular interest here whether there are particularly successful therapeutic strategies depending on gender and diagnosis with regard to the above-mentioned outcome parameters, i.e. whether there is a need to treat women and men differently if, for example, the tumor characteristics have the same tumor characteristics.

Since both analyses complement each other in their statements, the project can thus provide a comprehensive picture of gender-specific care in Germany. Furthermore, the project results provide a scientific data basis for a possible revision of the S3 guideline for the treatment of gastric cancer as well as for medical education and training.

ELIGIBILITY:
Inclusion Criteria:

Gastric adenocarcinoma ICD-10-GM code C16, C16.1 - C16.9

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A) Cases from the DRG statistics for the years 2017-2021 with inclusion criteria minimum age 18 years, full inpatient hospital treatment in the years 2017-2021, ICD-10-GM code C16, C16.1 - C16.9 B) Cases recorded in a clinical cancer registry from 2017-2021 with ICD-10-GM code C16, C16.1-C16.9
Sampling Method: Non-Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
DRG statistic: in-hospital mortality | 2017-2021
  Death in hospital after treatment in days
Cancer registry: 1 and 3 year survival | 2017-2021
  Survival after diagnosis date in months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School Brandenburg, Brandenburg, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: No
Due to data protection

REFERENCES:
- [Derived] Weber U, Kress L, Hunger R, Schildberg C, Mantke R. Gender differences in gastric cancer care and its adherence to guidelines in Germany (MaGen): protocol for an observational retrospective cohort study with administrative routine and cancer registry data from 2017 to 2021. BMJ Open. 2026 Feb 2;16(2):e103467. doi: 10.1136/bmjopen-2025-103467. PMID 41628928